CLINICAL TRIAL: NCT06239454
Title: Interleaving Stimulation Improves Dyskinesia in Parkinson's Disease: Randomized, Double-blind, Controlled Trial
Brief Title: Interleaving Stimulation Improves Dyskinesia in Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huashan Hospital (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Jian Wang, Professor of neuroloy department, Huashan Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KY2022-507
Record Dates: First submitted 2023-12-14; First posted 2024-02-02 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Parkinson's Disease
Keywords: Interleaving stimulation; dyskinesia syndrome in in Parkinson's disease; randomized, double-blind, controlled trial
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: 50 Patients will be randomly assigned to either the interleaving stimulation modes group (ISG) or the empirical stimulation modes group (ESG).
  ISG: empirical stimulation for the first 3 months, followed by interleaving programming period for 6 months, and any stimulation decided by the neurologists/neurosurgeons for the final 3 months.
  ESG: empirical programming for the first 9 months' period, followed by any stimulation decided by the neurologists/neurosurgeons for the final 3 months.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Randomization is done by computer-generated pairwise according to order of enrolment, so that similar numbers of patients are recruited to each study group. The chief investigator generates the randomization sequence. The randomization scheme is kept in sealed envelopes. The randomization sequence was revealed only to the unmasked clinician responsible for the stimulation programming, but not to the rater. Patients were masked to randomisation group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- empirical stimulation modes group (ESG) (Active Comparator): empirical programming for the first 9 months' period, followed by any stimulation decided by the neurologists/neurosurgeons for the final 3 months.
  Interventions: Device: empirical stimulation
- interleaving stimulation modes group (ISG) (Experimental): empirical stimulation for the first 3 months, followed by interleaving programming period for 6 months, and any stimulation decided by the neurologists/neurosurgeons for the final 3 months.
  Interventions: Device: interleaving stimulation

INTERVENTIONS:
Device: interleaving stimulation — ILS consists of two rapid and alternate stimulation programs with different contacts, amplitudes, and pulse width but the same frequency up to a maximum of 125Hz. Contact selection is determined by postoperative stereotactic computed tomography and clinical evaluation to achieve a balance between motor improvement and tolerable side effects. For example, ILS is successfully applied for PD motor symptoms (stimulation of subthalamic nucleus) as well as dyskinesia (additional stimulation of zona incerta).
  Arms: interleaving stimulation modes group (ISG)
Device: empirical stimulation — Patients are settled with simple polar stimulation with combined parameters adjustment (monopolar mode, 60~90µs pulse width, 130~185Hz frequency and varied voltage) during the follow-up.
  Arms: empirical stimulation modes group (ESG)

SUMMARY:
This study is designed as a prospective, randomized, double-blind, controlled study to assess putative differences in the effect of interleaving stimulation and empirical stimulation with regards to post-operation dyskinesia control. The primary objective is to assess putative differences in the effect of interleaving stimulation and empirical stimulation with regards to dyskinesia control.

DETAILED DESCRIPTION:
This study is designed as a prospective, randomized, double-blind, controlled study to assess putative differences in the effect of interleaving stimulation and empirical stimulation with regards to post-operation dyskinesia control. The primary objective is to assess putative differences in the effect of interleaving stimulation and empirical stimulation with regards to dyskinesia control.

50 Patients will be randomly assigned to either the interleaving stimulation modes group (ISG) or the empirical stimulation modes group (ESG). In ISG, empirical stimulation for the first 3 months, followed by interleaving programming period for 6 months, and any stimulation decided by the neurologists/neurosurgeons for the final 3 months. In ESG, empirical programming for the first 9 months' period, followed by any stimulation decided by the neurologists/neurosurgeons for the final 3 months. The change of dyskinesia scores (UPDRS IV, item 32 + item 33), Parkinson's disease quality of life-39 (PDQ-39) scores, scores of United Parkinson's Disease Rating Scale Part III as well as scores of neuropsychological Battery in interleaving stimulation compared to empirical programming modes will be measured based on corresponding time frame. Finally, the results will be analyzed via proper statistical methods and thus the conclusion will be drawn.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients at the age of 30-65 years old. 2. Patients diagnosed as Parkinson's disease according to the UK Parkinson's Disease Society Brain Bank criteria.

  3. Patients at Hoehn and Yahr stage 3 or lower in the on-state and stage 2 - 4 in the off-state.

  4. The disease duration of 5 years or more. 5. Patients with deep levodopa-responsive Parkinson's disease, and are not adequately controlled by drug therapy.

Exclusion Criteria:

* major illness or medical comorbidities, depression that is untreated but judged to be clinically significant by an investigator, cochlear implants, cardiac pacemakers, needs for diathermy, anticoagulant therapy, previous neuro-surgical procedure or ablative therapy, frank dementia according to cognitive screening, drug or alcohol abuse, being a woman of child-bearing potential, having a positive pregnancy test, or presence of a terminal illness.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
dyskinesia scores (United Parkinson's Disease Rating Scale Part IV, item 32 + item 33) | 3 months and 9 months
  Measure the changes of dyskinesia scores (United Parkinson's Disease Rating Scale Part IV, item 32 + item 33) in interleaving stimulation compared to empirical programming modes. The total scores range from 0 (good health) to 4 (poor health).
Parkinson's disease quality of life-39 (PDQ-39) scores | 3 months and 9 months
  Measure the changes of Parkinson's disease quality of life-39 (PDQ-39) scores in interleaving stimulation compared to empirical programming modes. The total scores range from 0 (good health) to 156 (poor health).

SECONDARY OUTCOMES:
scores of United Parkinson's Disease Rating Scale Part III | 3 months and 9 months
  Measure the changes of scores of United Parkinson's Disease Rating Scale Part III in interleaving stimulation compared to empirical programming modes. The total scores range from 0 (good health) to 132 (poor health).
Montreal cognitive assessment scores | 3 months and 9 months
  Measure the scores of Montreal cognitive assessment in interleaving stimulation compared to empirical programming modes. The total scores range from 0 (poor cognition) to 30 (good cognition).

CONTACTS AND LOCATIONS:
Overall Officials: Feng-Tao Liu, MD, Study Director — Huashan Hospital
Locations (1):
- Huashan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wiens BL, Iglewicz B. Design and analysis of three treatment equivalence trials. Control Clin Trials. 2000 Apr;21(2):127-37. doi: 10.1016/s0197-2456(99)00052-5. PMID 10715510
- [Background] Schuepbach WM, Rau J, Knudsen K, Volkmann J, Krack P, Timmermann L, Halbig TD, Hesekamp H, Navarro SM, Meier N, Falk D, Mehdorn M, Paschen S, Maarouf M, Barbe MT, Fink GR, Kupsch A, Gruber D, Schneider GH, Seigneuret E, Kistner A, Chaynes P, Ory-Magne F, Brefel Courbon C, Vesper J, Schnitzler A, Wojtecki L, Houeto JL, Bataille B, Maltete D, Damier P, Raoul S, Sixel-Doering F, Hellwig D, Gharabaghi A, Kruger R, Pinsker MO, Amtage F, Regis JM, Witjas T, Thobois S, Mertens P, Kloss M, Hartmann A, Oertel WH, Post B, Speelman H, Agid Y, Schade-Brittinger C, Deuschl G; EARLYSTIM Study Group. Neurostimulation for Parkinson's disease with early motor complications. N Engl J Med. 2013 Feb 14;368(7):610-22. doi: 10.1056/NEJMoa1205158. PMID 23406026
- [Background] Odekerken VJ, van Laar T, Staal MJ, Mosch A, Hoffmann CF, Nijssen PC, Beute GN, van Vugt JP, Lenders MW, Contarino MF, Mink MS, Bour LJ, van den Munckhof P, Schmand BA, de Haan RJ, Schuurman PR, de Bie RM. Subthalamic nucleus versus globus pallidus bilateral deep brain stimulation for advanced Parkinson's disease (NSTAPS study): a randomised controlled trial. Lancet Neurol. 2013 Jan;12(1):37-44. doi: 10.1016/S1474-4422(12)70264-8. Epub 2012 Nov 16. PMID 23168021
- [Background] Koeglsperger T, Palleis C, Hell F, Mehrkens JH, Botzel K. Deep Brain Stimulation Programming for Movement Disorders: Current Concepts and Evidence-Based Strategies. Front Neurol. 2019 May 21;10:410. doi: 10.3389/fneur.2019.00410. eCollection 2019. PMID 31231293
- [Background] Kern DS, Picillo M, Thompson JA, Sammartino F, di Biase L, Munhoz RP, Fasano A. Interleaving Stimulation in Parkinson's Disease, Tremor, and Dystonia. Stereotact Funct Neurosurg. 2018;96(6):379-391. doi: 10.1159/000494983. Epub 2019 Jan 17. PMID 30654368
- [Background] Zhang S, Zhou P, Jiang S, Wang W, Li P. Interleaving subthalamic nucleus deep brain stimulation to avoid side effects while achieving satisfactory motor benefits in Parkinson disease: A report of 12 cases. Medicine (Baltimore). 2016 Dec;95(49):e5575. doi: 10.1097/MD.0000000000005575. PMID 27930569
- [Background] Franca C, Barbosa ER, Iglesio R, Teixeira MJ, Cury RG. Interleaving Stimulation in Parkinson Disease: Interesting to Whom? World Neurosurg. 2019 Oct;130:e786-e793. doi: 10.1016/j.wneu.2019.06.223. Epub 2019 Jul 8. PMID 31295615
- [Background] Khabarova EA, Denisova NP, Dmitriev AB, Slavin KV, Verhagen Metman L. Deep Brain Stimulation of the Subthalamic Nucleus in Patients with Parkinson Disease with Prior Pallidotomy or Thalamotomy. Brain Sci. 2018 Apr 16;8(4):66. doi: 10.3390/brainsci8040066. PMID 29659494
- [Background] Bouthour W, Bereau M, Kibleur A, Zacharia A, Tomkova Chaoui E, Fleury V, Benis D, Momjian S, Bally J, Luscher C, Krack P, Burkhard PR. Dyskinesia-inducing lead contacts optimize outcome of subthalamic stimulation in Parkinson's disease. Mov Disord. 2019 Nov;34(11):1728-1734. doi: 10.1002/mds.27853. Epub 2019 Sep 30. PMID 31571277
- [Background] Picillo M, Lozano AM, Kou N, Puppi Munhoz R, Fasano A. Programming Deep Brain Stimulation for Parkinson's Disease: The Toronto Western Hospital Algorithms. Brain Stimul. 2016 May-Jun;9(3):425-437. doi: 10.1016/j.brs.2016.02.004. Epub 2016 Feb 12. PMID 26968806
- [Background] Aquino CC, Duffley G, Hedges DM, Vorwerk J, House PA, Ferraz HB, Rolston JD, Butson CR, Schrock LE. Interleaved deep brain stimulation for dyskinesia management in Parkinson's disease. Mov Disord. 2019 Nov;34(11):1722-1727. doi: 10.1002/mds.27839. Epub 2019 Sep 4. PMID 31483534
- See also: Devroye, Luc. 1986. Non-Uniform Random Variate Generation. Springer-Verlag. New York. — https://link.springer.com/book/10.1007/978-1-4613-8643-8

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-05-20): https://cdn.clinicaltrials.gov/large-docs/54/NCT06239454/Prot_SAP_000.pdf
  • Informed Consent Form (2022-05-20): https://cdn.clinicaltrials.gov/large-docs/54/NCT06239454/ICF_001.pdf